CLINICAL TRIAL: NCT02460198
Title: A Phase II Study of Pembrolizumab (MK-3475) as Monotherapy in Subjects With Previously Treated Locally Advanced Unresectable or Metastatic (Stage IV) Mismatched Repair Deficient or Microsatellite Instability-High Colorectal Carcinoma (KEYNOTE-164)
Brief Title: Study of Pembrolizumab (MK-3475) as Monotherapy in Participants With Previously-Treated Locally Advanced Unresectable or Metastatic Colorectal Cancer (MK-3475-164/KEYNOTE-164)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-164; 153046 (Registry Identifier: JAPIC-CTI); MK-3475-164 (Other: Merck Protocol Number); KEYNOTE-164 (Other: Merck); 2015-001852-32 (EudraCT Number)
Record Dates: First submitted 2015-05-29; First posted 2015-06-02 (Estimated); Results first posted 2020-08-21 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Carcinoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); MSI-H; MSI
MeSH Terms: conditions — Colorectal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A - Pembrolizumab 200 mg (Experimental): Participants were previously treated with standard therapies, which must include fluoropyrimidine, oxaliplatin, and irinotecan. Cohort A participants receive pembrolizumab 200 mg intravenously (IV) on Day 1 of every 3-week cycle (Q3W) for up to approximately 52 cycles (up to approximately 3 years).
  Interventions: Biological: Pembrolizumab
- Cohort B - Pembrolizumab 200 mg (Experimental): Participants were previously treated with at least one line of systemic standard of care therapy: fluoropyrimidine + oxaliplatin or fluoropyrimidine + irinotecan +/ - anti vascular endothelial growth factor (VEGF)/ epidermal growth factor regulator (EGFR) monoclonal antibody. Cohort B participants receive pembrolizumab 200 mg IV on Day 1 Q3W for up to approximately 52 cycles (up to approximately 3 years).
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®

SUMMARY:
In this study, participants with previously-treated locally-advanced unresectable or metastatic mismatched repair (MMR) deficient or microsatellite instability-high (MSI-H) colorectal carcinoma (CRC) will be treated with pembrolizumab (MK-3475, KEYTRUDA®) monotherapy.

There will be two cohorts in this study: Cohort A and Cohort B. For Cohort A, participants are required to have been previously treated with standard therapies, which must include fluoropyrimidine, oxaliplatin, and irinotecan. Enrollment into Cohort A has been completed. For Cohort B, participants are required to have been previously treated with at least one line of systemic standard of care therapy: fluoropyrimidine + oxaliplatin or fluoropyrimidine + irinotecan +/ - anti-vascular endothelial growth factor (VEGF)/ epidermal growth factor regulator (EGFR) monoclonal antibody.

The primary hypothesis is that Objective Response Rate (ORR) based on Response Evaluation Criteria in Solid Tumors v 1.1 (RECIST 1.1) assessed by central imaging vendor in participants with locally advanced unresectable or metastatic MMR deficient or MSI high CRC is greater than 15%.

DETAILED DESCRIPTION:
With protocol amendment 08 (13-Nov-2019), once study participants have achieved the study objective or the study has ended, participants will be discontinued from this study and may be enrolled in a pembrolizumab extension study (NCT03486873) to continue protocol-defined assessments and treatment.

ELIGIBILITY:
Inclusion criteria:

* Histologically-proven locally advanced unresectable or metastatic colorectal carcinoma
* Locally confirmed MMR deficient or MSI-H status
* Has been previously treated with standard therapies, which must include, for Cohort A, fluoropyrimidine, oxaliplatin, and irinotecan, and for Cohort B, at least one line of systemic standard of care therapy: fluoropyrimidine + oxaliplatin or fluoropyrimidine + irinotecan +/- anti-VEGF/EGFR monoclonal antibody (mAb).
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Life expectancy of greater than 3 months
* Provides an archival or newly obtained (≤60 days prior to first dose of study treatment) tumor tissue sample (Cohort B)
* At least one measurable lesion
* Female participants of childbearing potential should be willing to use acceptable methods of contraception or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study treatment
* Male participants should agree to use an adequate method of contraception starting with the first dose of study treatment through 120 days after the last dose of study treatment
* Adequate organ function

Exclusion criteria:

* Currently participating in another study and receiving trial treatment, participated in a study of an investigational agent and received trial treatment within 4 weeks of the first dose of treatment in this study, or used an investigational device within 4 weeks of the first dose of treatment in this study
* Active autoimmune disease that has required systemic treatment in past 2 years
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Known active central nervous system metastases and/or carcinomatous meningitis
* Prior monoclonal antibody (mAb), chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events (AEs) due to a previously administered agent
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Received a live vaccine within 30 days of planned start of study treatment
* Known history of human immunodeficiency virus (HIV)
* Known active Hepatitis B or C
* Has known history of, or any evidence of interstitial lung disease or active, noninfectious pneumonitis
* Active infection requiring systemic therapy
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-08-25 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2021-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Le DT, Kim TW, Van Cutsem E, Geva R, Jager D, Hara H, Burge M, O'Neil B, Kavan P, Yoshino T, Guimbaud R, Taniguchi H, Elez E, Al-Batran SE, Boland PM, Crocenzi T, Atreya CE, Cui Y, Dai T, Marinello P, Diaz LA Jr, Andre T. Phase II Open-Label Study of Pembrolizumab in Treatment-Refractory, Microsatellite Instability-High/Mismatch Repair-Deficient Metastatic Colorectal Cancer: KEYNOTE-164. J Clin Oncol. 2020 Jan 1;38(1):11-19. doi: 10.1200/JCO.19.02107. Epub 2019 Nov 14. PMID 31725351
- [Result] Le DT, Diaz LA Jr, Kim TW, Van Cutsem E, Geva R, Jager D, Hara H, Burge M, O'Neil BH, Kavan P, Yoshino T, Guimbaud R, Taniguchi H, Elez E, Al-Batran SE, Boland PM, Cui Y, Leconte P, Marinello P, Andre T. Pembrolizumab for previously treated, microsatellite instability-high/mismatch repair-deficient advanced colorectal cancer: final analysis of KEYNOTE-164. Eur J Cancer. 2023 Jun;186:185-195. doi: 10.1016/j.ejca.2023.02.016. Epub 2023 Feb 24. PMID 37141828
- [Derived] van Vugt MJH, Stone JA, De Greef RHJMM, Snyder ES, Lipka L, Turner DC, Chain A, Lala M, Li M, Robey SH, Kondic AG, De Alwis D, Mayawala K, Jain L, Freshwater T. Immunogenicity of pembrolizumab in patients with advanced tumors. J Immunother Cancer. 2019 Aug 8;7(1):212. doi: 10.1186/s40425-019-0663-4. PMID 31395089
- See also: Merck Clinical Trials Information — https://merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 34 clinical sites in 10 countries.
Pre-assignment Details: Participant flow as per the database cutoff date of 19FEB2021.
Groups:
- Cohort A - Pembrolizumab 200 mg: Participants were previously treated with standard therapies, which included fluoropyrimidine, oxaliplatin, and irinotecan. Cohort A participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of every 3-week cycle (Q3W) for up to approximately 52 cycles (up to approximately 3 years), which included a first course of 35 cycles and second course treatment phase of 17 cycles after experiencing PD if criteria were met for re-treatment.
- Cohort B - Pembrolizumab 200 mg: Participants were previously treated with at least one line of systemic standard of care therapy: fluoropyrimidine + oxaliplatin or fluoropyrimidine + irinotecan +/ - anti vascular endothelial growth factor (VEGF)/ epidermal growth factor regulator (EGFR) monoclonal antibody. Cohort B participants received pembrolizumab 200 mg IV on Day 1 Q3W for up to approximately 52 cycles (up to approximately 3 years), which included a first course of 35 cycles and second course treatment phase of 17 cycles after experiencing PD if criteria were met for re-treatment.
Period: Overall Study
Arm/Group | Cohort A - Pembrolizumab 200 mg | Cohort B - Pembrolizumab 200 mg
Started | 61 | 63
Completed | 0 | 0
Not Completed | 61 | 63
Not completed — Adverse Event | 1 | 3
Not completed — Death | 36 | 28
Not completed — Lost to Follow-up | 1 | 1
Not completed — Transferred to Extension Study | 15 | 15
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Site Terminated By Sponsor | 0 | 1
Not completed — Did Not Continue on Extension Study | 6 | 11

BASELINE CHARACTERISTICS:
Population: The analysis population included all randomized and treated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A - Pembrolizumab 200 mg | Cohort B - Pembrolizumab 200 mg | Total
Number analyzed (Participants) | 61 | 63 | 124
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.3 (14.5) | 57.8 (15.2) | 56.1 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 30 | 55
  Male | 36 | 33 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 59 | 60 | 119
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 19 | 14 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 7 | 7
  White | 42 | 42 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) - Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) Assessed by Central Imaging Vendor
Description: Objective response rate was defined as the percentage of the participants in the analysis population who had a complete response (CR) or partial response (PR). Complete Response: disappearance of all target lesions. Partial Response: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Responses were based upon blinded central imaging vendor per RECIST 1.1. The point estimate and 95% confidence interval for the ORR, were provided using an exact binomial distribution (Clopper and Pearson method). Participants without response data were counted as nonresponders. The data cutoff date was 09-SEPT-2019.
Time Frame: Up to approximately 48 months
Population: The analysis population consisted of all participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Cohort A - Pembrolizumab 200 mg: Participants were previously treated with standard therapies, which must include fluoropyrimidine, oxaliplatin, and irinotecan. Cohort A participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of every 3-week cycle (Q3W) for up to approximately 35 cycles (up to approximately 2 years).
- Cohort B - Pembrolizumab 200 mg: Participants were previously treated with at least one line of systemic standard of care therapy: fluoropyrimidine + oxaliplatin or fluoropyrimidine + irinotecan +/ - anti vascular endothelial growth factor (VEGF)/ epidermal growth factor regulator (EGFR) monoclonal antibody. Cohort B participants received pembrolizumab 200 mg IV on Day 1 Q3W for up to approximately 35 cycles (up to approximately 2 years).
Arm/Group | Cohort A - Pembrolizumab 200 mg | Cohort B - Pembrolizumab 200 mg
Number analyzed (Participants) | 61 | 63
Percentage of participants | 32.8 [21.3 to 46.0] | 34.9 [23.3 to 48.0]

2. Secondary Outcome: Disease Control Rate (DCR) Per RECIST 1.1 Assessed by Central Imaging Vendor.
Description: Disease Control Rate was defined as the percentage of participants who achieved confirmed CR or PR or had demonstrated stable disease (SD) for at least 24 weeks prior to any evidence of progression. Complete Response: disappearance of all target lesions. Partial Response: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease: neither sufﬁcient shrinkage to qualify for PR nor sufﬁcient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study. Progressive Disease: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. or the appearance of new lesion(s). Participants in the analysis population with missing DCR were considered as disease not under control. The data cutoff date was 19-Feb-2021.
Time Frame: Up to approximately 66 months
Population: The analysis population consisted of all participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A - Pembrolizumab 200 mg | Cohort B - Pembrolizumab 200 mg
Number analyzed (Participants) | 61 | 63
Percentage of participants | 50.8 [37.7 to 63.9] | 55.6 [42.5 to 68.1]

3. Secondary Outcome: Progression-Free Survival (PFS) Per RECIST 1.1 Assessed by Central Imaging Vendor.
Description: PFS is defined as the time from first day of study treatment to the first documented disease progression or death due to any cause, whichever occurs first. Progressive Disease: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions was also considered progression). PFS was summarized by Kaplan-Meier (KM) methods. The data cutoff date was 19-FEB-2021.
Time Frame: Up to approximately 66 months
Population: The analysis population consisted of all participants who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A - Pembrolizumab 200 mg | Cohort B - Pembrolizumab 200 mg
Number analyzed (Participants) | 61 | 63
Months | 2.3 [2.1 to 8.1] | 4.1 [2.1 to 18.9]

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from first day of study treatment to death due to any cause. Participants without documented death at the time of analysis are censored at the date of the last follow-up. OS was summarized by Kaplan-Meier (KM) methods. The data cutoff date was 19-FEB-2021.
Time Frame: Up to approximately 66 months
Population: The analysis population consisted of all participants who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A - Pembrolizumab 200 mg | Cohort B - Pembrolizumab 200 mg
Number analyzed (Participants) | 61 | 63
Months | 31.4 [21.4 to 58] | 47 [19.2 to NA] — NA = OS upper limit was not reached (insufficient number of deaths by time of last disease assessment).

5. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE).
Description: An adverse event (AE) was defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it was considered related to the medical treatment or procedure, that occurred during the course of the study.
Time Frame: Up to approximately 66 months
Population: The analysis population consisted of all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A - Pembrolizumab 200 mg | Cohort B - Pembrolizumab 200 mg
Number analyzed (Participants) | 61 | 63
Participants | 60 | 63

6. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE.
Description: as for outcome 5
Time Frame: Up to approximately 36 months
Population: The analysis population consisted of all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A - Pembrolizumab 200 mg | Cohort B - Pembrolizumab 200 mg
Number analyzed (Participants) | 61 | 63
Participants | 5 | 5

7. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 as Assessed by the Central Imaging Vendor
Description: For participants who demonstrated a CR or PR, duration of response was defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurred first. Complete Response: disappearance of all target lesions. Partial Response: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Responses were based upon blinded central imaging vendor per RECIST 1.1. Duration of Response was based on Independent radiologist review (IRC) using RECIST 1.1 and was summarized by Kaplan-Meier (KM) methods for censored data. Nonresponders were excluded from the analysis of DOR.
Time Frame: Up to approximately 66 months
Population: The analysis population consisted of all participants who received at least one dose of study treatment and demonstrated a CR or PR.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A - Pembrolizumab 200 mg | Cohort B - Pembrolizumab 200 mg
Number analyzed (Participants) | 20 | 22
Months | NA [6.2 to NA] — NA = Median DOR and DOR upper limit were not reached by the time of last disease assessment. | NA [4.4 to NA] — NA = Median DOR and DOR upper limit were not reached by the time of last disease assessment.

ADVERSE EVENTS:
Time Frame: Up to approximately 66 months
Description: Adverse events were collected for a minimum of 30 days after the end of treatment and every 12 weeks during follow-up. The analysis population for AEs included all randomized participants who received at least one dose of study medication whereas the analysis population for deaths included all randomized participants. MedDRA preferred terms "Neoplasm Progression", "Malignant Neoplasm Progression", and "Disease Progression" not related to the drug were excluded. Database Cutoff Date: 19FEB2021
Groups:
- Cohort A First Course: Participants were previously treated with standard therapies, which must include fluoropyrimidine, oxaliplatin, and irinotecan. Cohort A participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of every 3-week cycle (Q3W) for up to approximately 35 cycles (up to approximately 2 years).
- Cohort B First Course: Participants were previously treated with at least one line of systemic standard of care therapy: fluoropyrimidine + oxaliplatin or fluoropyrimidine + irinotecan +/ - anti vascular endothelial growth factor (VEGF)/ epidermal growth factor regulator (EGFR) monoclonal antibody. Cohort B participants received pembrolizumab 200 mg IV on Day 1 Q3W for up to approximately 35 cycles (up to approximately 2 years).
- Cohort A Second Course; Cohort B Second Course: Participants who completed first course of treatment were treated with pembrolizumab 200 mg intravenously (IV) on Day 1 of every 3-week cycle (Q3W) for up to 17 cycles (approximately 1 year) after experiencing PD if criteria were met for re-treatment.
Arm/Group | Cohort A First Course | Cohort B First Course | Cohort A Second Course | Cohort B Second Course
All-Cause Mortality (participants affected / at risk) | 38/61 | 31/63 | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 31/61 | 25/63 | 1/6 | 1/3
Other Adverse Events (participants affected / at risk) | 56/61 | 58/63 | 5/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A First Course (N=61) | Cohort B First Course (N=63) | Cohort A Second Course (N=6) | Cohort B Second Course (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal decompensation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 3 (7) | 0 (0) | 0 (0) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (5) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Euthanasia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Biloma (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alkalosis hypochloraemic (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autoimmune arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscle swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A First Course (N=61) | Cohort B First Course (N=63) | Cohort A Second Course (N=6) | Cohort B Second Course (N=3)
Anaemia (Blood and lymphatic system disorders) | 12 (21) | 11 (13) | 2 (4) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 4 (5) | 7 (7) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 6 (6) | 13 (15) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 18 (26) | 14 (18) | 1 (1) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 13 (15) | 13 (14) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 23 (46) | 16 (28) | 1 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 5 (7) | 9 (9) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 22 (32) | 17 (26) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 2 (3) | 2 (3) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 3 (5) | 0 (0) | 1 (2)
Toothache (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 18 (37) | 14 (18) | 1 (2) | 0 (0)
Asthenia (General disorders) | 14 (20) | 5 (6) | 0 (0) | 0 (0)
Chills (General disorders) | 3 (4) | 4 (4) | 0 (0) | 0 (0)
Fatigue (General disorders) | 19 (24) | 24 (29) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 4 (5) | 7 (11) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 11 (12) | 10 (10) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 13 (22) | 11 (19) | 2 (5) | 0 (0)
Conjunctivitis (Infections and infestations) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (9) | 2 (2) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 4 (8) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 8 (13) | 8 (10) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (7) | 5 (7) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Stoma site pruritus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 8 (11) | 7 (10) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 6 (9) | 5 (7) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 5 (7) | 3 (5) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 7 (7) | 1 (1) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 14 (16) | 11 (13) | 2 (3) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 6 (7) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (5) | 4 (14) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (12) | 3 (3) | 1 (1) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (26) | 16 (19) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 14 (18) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (9) | 3 (3) | 1 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 7 (7) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (8) | 0 (0) | 1 (2)
Amnesia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5) | 3 (3) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (4) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 9 (11) | 8 (16) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 4 (6) | 2 (2) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (4) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (3) | 5 (5) | 1 (1) | 0 (0)
Drug dependence (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 8 (8) | 5 (6) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (5) | 2 (2) | 1 (2) | 0 (0)
Urinary tract discomfort (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (20) | 9 (9) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 8 (9) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (8) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (15) | 8 (9) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 8 (13) | 9 (18) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5) | 0 (0) | 0 (0)
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 5 (9) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.

Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT02460198/Prot_SAP_001.pdf